CLINICAL TRIAL: NCT01356615
Title: Low Molecular Weight Heparin (Enoxaparin Sodium) and Standard Unfractionated Heparin for Hemodialysis Anticoagulation
Brief Title: Low Molecular Weight Heparin for Hemodialysis Anticoagulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Mahboob Lessan-Pezeshki, Department of Nephrology and Dialysis, Imam Khomeini Hospital. Tehran University of Medical Sciences, Tehran, Iran
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 814; enoxaparin sodium and UFH (Other: Tehran University of Medical Sciences)
Record Dates: First submitted 2011-04-15; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: anticoagulation; hemodialysis; heparin; lipids; low molecular weight heparins
MeSH Terms: interventions — Heparin, Low-Molecular-Weight; enoxaparin sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- enoxaparin (Experimental): enoxaparin sodium (Clexane) (40 mg) followed prospectively for 3 months (36 dialyses)
  Interventions: Drug: low molecular weight heparin (enoxaparin sodium)
- standard unfractionated heparin (Active Comparator): standard unfractionated heparin followed prospectively for 3 months (36 dialyses)
  Interventions: Drug: standard unfractionated heparin

INTERVENTIONS:
Drug: low molecular weight heparin (enoxaparin sodium) — Enoxaparin sodium (Clexane; 40 mg) was administered 3-4 min before dialysis as a bolus dose, into the arterial line pre-dialyzer.
  Arms: enoxaparin
Drug: standard unfractionated heparin — Heparin (sodium heparin 5000 IU/ml) was administered as a bolus dose (50 IU/kg body weight) intravenously into the pre-dialyzer arterial line of the extracorporeal blood circuit, followed by a maintenance dose of 1000 IU sodium heparin per hour.
  Arms: standard unfractionated heparin

SUMMARY:
Low-molecular weight heparins (LMWHs) as well as Unfractionated heparin (UFH) is used as anticoagulation during hemodialysis (HD) therapy. In this study the investigators have compared clinical efficacy and safety of LMWH and UFH, and their effect on lipid profile.

DETAILED DESCRIPTION:
In this prospective, randomized, cross-over study the investigators compared the safety, clinical efficacy of Clexane (enoxaparin sodium; Sanofi-Aventis) with unfractionated heparin in 27 chronic HD patients. Group A received Clexane (enoxaparin sodium; Sanofi-Aventis) and were followed up for 3 months and then crossed over to Unfractionated heparin for a further 3-month period. Group B received Unfractionated heparin first and then crossed over to Clexane, each followed up for 3 months. Heparin anticoagulation, clinical clotting and hemorrhage were evaluated by visual inspection after blood draining of the air trap.

ELIGIBILITY:
Inclusion Criteria:

* patients in end stage renal failure requiring maintenance dialysis were recruited into the study

Exclusion Criteria:

* Patients with known bleeding disorders
* Subjects receiving oral or other forms of anticoagulant therapy (e.g. warfarin, aspirin) or drugs that could affect heparin activity (e.g. digitalis, tetracyclines, and antihistamines) were also excluded. Subjects continued their usual medication (including lipid-lowering therapy ) and were treated in the normal manner by their caring physicians during the study.

Ages: 25 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Fibrin/clot formation in the dialyzer and Hemorrhage in Dialysis by visual inspection | 3 month
  The frequency and degree of clot and fibrin formation in both the dialyzer and lines were scored on a 10-point scale, with 1 indicating no clot formation and 10 sever clotting or total occlusion. This assessment was done after the blood had been returned to the patient by flushing the dialyzer and lines with normal saline. Hemorrhage or thrombosis, during and between dialyses was also noted. Heparin anticoagulation, Clinical clotting and Hemorrhage were evaluated by visual inspection.
  Hemorrhages were categorized as weak, moderate, and severe.

SECONDARY OUTCOMES:
changes in serum Cholesterol,low and High Density Lipoprotein and Triglycerid. | 3 month
  27 chronic HD patients. They were randomly assigned to either Clexane (40 mg) or standard heparin, and followed prospectively for 3 months (36 dialyses) and then crossed over to the alternate therapy for a further 3 months Fasting standard lipid profiles were determined at the end of each arm of the study. Total cholesterol (TC), high density lipoprotein (HDL), and triglyceride (TG) were measured.

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593